CLINICAL TRIAL: NCT01620515
Title: Phase 2 Multicenter Prospective Open Label 2-Dose Level Clinical Safety and Efficacy Evaluation of Injection of NX-1207 for the Treatment of Low Risk, Localized (T1c) Prostate Cancer
Brief Title: Two-Dose Level Evaluation of NX-1207 for the Treatment of Low Risk, Localized (T1c) Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nymox Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NX03-0040
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Prostate Cancer
Keywords: Prostate; Prostate Cancer; Localized Prostate Cancer; T1c Prostate Cancer; Focal Therapy; NX-1207
MeSH Terms: conditions — Prostatic Neoplasms | interventions — fexapotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Active Surveillance (No Intervention): Subjects with low risk localized (T1c) prostate cancer who are being followed with active surveillance and not undergoing active treatment for prostate cancer.
- NX-1207 2.5 mg (Experimental)
  Interventions: Drug: NX-1207 2.5 mg
- NX-1207 15 mg (Experimental)
  Interventions: Drug: NX-1207 15 mg

INTERVENTIONS:
Drug: NX-1207 2.5 mg — A single intraprostatic injection of NX-1207 2.5 mg followed by active surveillance.
  Arms: NX-1207 2.5 mg
Drug: NX-1207 15 mg — A single intraprostatic injection of NX-1207 15 mg followed by active surveillance.
  Arms: NX-1207 15 mg

SUMMARY:
This study is designed to evaluate the safety and efficacy of a single injection of NX-1207 for the treatment of biopsy-confirmed low risk localized (T1c) prostate cancer in patients currently undergoing active surveillance. Study participants currently on active surveillance will be randomized either to treatment with a single intraprostatic injection of NX-1207 (2.5 mg or 15 mg) followed by active surveillance or to no treatment (continued active surveillance). Blinded efficacy evaluation will be by a second post-treatment prostate biopsy.

ELIGIBILITY:
Inclusion Criteria:

* T1c prostate cancer
* Gleason score ≤ 6 with no Gleason pattern of 4 or 5.
* Life expectancy ≥ 5 years.
* Single positive prostate biopsy core with ≤ 50% cancer
* PSA ≤ 10 ng/mL

Exclusion Criteria:

* Previous active treatment (such as surgery, brachytherapy, radiotherapy) for prostate cancer.
* Evidence of metastatic disease or previous positive bone scan.
* Previous hormonal therapy for prostate cancer.
* Use of certain concomitant medications, including 5 alpha reductase inhibitors (e.g. finasteride, dutasteride), androgen receptor blockers (e.g. flutamide, bicalutamide), immunosuppressants(such as Imuran™, Enbrel™, Remicade™, Humira™, etc.), anticoagulants(such as Coumadin™ or heparin), or chemotherapeutics.
* Previous surgical or invasive prostate treatments such as TURP, TUMT, TUNA, laser or any other minimally invasive treatment within the past 12 months.
* Pelvic irradiation.
* Urinary tract infection more than once in the past 12 months.
* Acute or chronic prostatitis in the past 12 months.
* Clinically significant renal or hepatic impairment.
* Bleeding disorder.
* Poorly controlled diabetes type 1 or type 2.
* Urinary retention in the previous 12 months.
* Self-catheterization for urinary retention.
* Post-void residual urine volume > 200 mL.
* Prior significant rectal surgery or any rectal condition with rectal stenosis or fistula.
* History of alcohol or substance abuse or dependence within the past 2 years.

Ages: 45 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2012-02-21 (Actual); Primary Completion 2015-10-21 (Actual); Study Completion 2015-10-21 (Actual)

PRIMARY OUTCOMES:
Undetectable cancer post-treatment in the region of the prostate where the baseline cancer was detected. | Baseline to 45 days post-treatment
  The primary efficacy endpoint is the percentage of subjects with undetectable prostate cancer (negative biopsy) in the region of the prostate where the baseline cancer was detected.
Safety of a single treatment of NX-1207 2.5 mg or NX-1207 15 mg in subjects with biopsy-confirmed low grade low risk localized (T1c) prostate cancer. | Baseline to 60 days post-treatment
  Safety will be assessed by physical exam, prostate biopsy, monitoring of adverse events, changes in ECG, and changes in PSA and other clinical laboratory values.

SECONDARY OUTCOMES:
Change in tumor grade in the region of the baseline prostate cancer | Baseline to 45 days post-treatment
Change in tumor volume in the region of the baseline prostate cancer | Baseline to 45 days post-treatment
Change in tumor grade for the whole prostate | Baseline to 45 days post-treatment
Change in tumor volume in the whole prostate | Baseline to 45 days post-treatment

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Tucson, Arizona
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Atherton, California
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., La Mesa, California
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Long Beach, California
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., San Diego, California
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Denver, Colorado
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Englewood, Colorado
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., New Britain, Connecticut
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Aventura, Florida
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Naples, Florida
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Jeffersonville, Indiana
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Shreveport, Louisiana
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Annapolis, Maryland
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Baltimore, Maryland
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Las Vegas, Nevada
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Brick, New Jersey
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Albuquerque, New Mexico
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Garden City, New York
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., New York, New York
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Myrtle Beach, South Carolina
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Germantown, Tennessee
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Carrollton, Texas
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Salt Lake City, Utah